| Official Title: | Randomized Comparison of Combination Azithromycin and Hydroxychloroquine vs. Hydroxychloroquine Alone for the Treatment of Confirmed COVID-19 |
|---|---|
| NCT number: | 04336332 |
| <b>Document Type:</b> | SAP |
| Date of the | 05/08/2020 |
| Document: | |

v

# 6.0 Data Management Plan

#### 6.1 Data Analysis

#### Statistical considerations

We follow Gautret et al. (2020) in using, as a primary endpoint, absence of viral evidence of disease six days following start of treatment. In that study (Table 3), there were 14 patients treated with hydroxychloroquine alone, and 8/14 (57.1 percent) of them were virus-free at 6 days. There were six patients treated with both hydroxychloroquine plus azithromycin, and all six (100%) were virus-free at 6 days. In a third group of patients with no hydroxychloroquine, there were 16 patients, of whom 2 (12.5 percent) were virus-free at 6 days.

We propose a three-arm trial as follows: Arm 1 (HCQ + AZ), Arm 2 (HCQ alone), and Arm 3 (delayed HCQ), with patients randomized 2:2:1. Arm 1 will be compared to Arm 2, and Arm 2 to Arm 3. A total of 160 patients will be accrued, with 60 patients in Arms 1 and 2 and 30 patients in Arm 3. The additional 10 patients accrued are to account for potential drop out of subjects. An interim analysis for futility will be carried out at the 50% target accrual point, which is after 75 patients have been enrolled. Randomization will be stratified on (A) in-patient vs out-patient, and (B) severe vs not severe, as defined in Section 1.3 to ensure that these factors are balanced among all three arms.

# HCQ + AZ versus HCQ alone

The primary outcome is a comparison of Arm 1 to Arm 2, with the aim of determining if the addition of AZ to HCQ is effective. The primary endpoint is the proportion of patients that are virus-free at 6 days. We assume that the proportion of patients in the hydroxychloroquine arm who are virus-free at 6 days is 0.571, and that the trial is stopped for futility at the 50% accrual point if the conditional power at that time is below 0.15. The following table shows the power of detecting an improvement in the outcome for a range of proportions virus-free in the combination arm.

| Proportion virus-free (HCQ only) | Proportion virus-<br>free HCQ plus | Proportion difference | Power no futility stopping | Loss of power with<br>futility stopping<br>(simulation) |
|---|---|---|---|---|
| 0.571 | 0.805 | 0.234 | 0.800 | 0.0019 |
| 0.571 | 0.820 | 0.249 | 0.851 | 0.0016 |
| 0.571 | 0.820 | 0.349 | 0.882 | 0.0013 |

For example, with 60 patients per arm, we could detect, with 80 percent power, an increase in the proportion of virus-free patients from 57.1 percent in the hydroxychloroquine arm to 80.5 percent in the combination arm. The loss of power associated with using futility stopping is only 0.19 percent.

The two-sided Type I error probability associated with this test is 0.05. We will use an uncorrected chi-squared statistic to evaluate this null hypothesis.

# HCQ versus placebo and delayed HCQ

A second, independent goal of the study is to ensure that, in fact, hydroxychloroquine is effective in reducing viral load. Thus, we plan a third, control arm, in which patients will receive a placebo for six days, at which time they will switch to receiving HCQ. We plan to compare Arms 2 and 3, with the

3) having 30 patients and the HCQ arm having 60 patients, as above. Based on the Gautret et al. study [9], we assume the baseline proportion of patients who are virus-free at six days is 0.125. The following table shows the detectable difference with a variety of baseline rates:

| Proportion virus-free<br>Control (delayed HCQ) | Proportion virus-<br>free HCQ | Proportion difference | Power no futility stopping | Loss of power with<br>futility stopping<br>(simulation) |
|---|---|---|---|---|
| 0.125 | 0.401 | 0.276 | 0.800 | 0.0005 |
| 0.125 | 0.420 | 0.249 | 0.848 | 0.0003 |
| 0.125 | 0.430 | 0.349 | 0.870 | 0.0005 |

Thus, for a range of plausible virus-free rates for the HCQ arm, the detectable rate for the HCQ arm is well within the range reported by Gautret et al [9]. The futility analysis has a negligible effect on power.

**Futility stopping rule** 

This clinical trial will use a non-binding futility stopping rule based on conditional power [20]. At the 50% accrual point (75 patients), an interim analysis will be carried out and the conditional power of the primary (Arm 1 vs Arm 2) and secondary (Arm 2 vs Arm 3) calculated. A data monitoring committee will review the analysis to determine if accrual to any of the arms should be stopped for futility.

Other analyses

A key secondary endpoint will be the number of days from initiation of therapy to VND (virtually no disease). This can be displayed graphically using Kaplan-Meier survival curves, and formally assessed using a log-rank test. Other secondary endpoints that can be assessed in this way are (1) Time in days to being afebrile for 48 hours, (2) time in days to resolution of symptoms (as assessed by a symptom questionnaire), (3) time in days to discharge (if hospitalized), (4) time to recovery (able to return to work or school), and (5) time to death from COVID-19. Other measures that will be assessed via descriptive statistics are agent toxicity, adverse events, and improvement over time in vital signs.

The effects of additional clinical variables on the primary outcome and other binary outcomes will be assessed via logistic regression. The effects of these variables on survival endpoints will be assessed via the Cox proportional hazards model. Numbers of patient deaths due to COVID-19 in the three arms will be compared using tests of proportions, and via log-rank test comparison of Kaplan-Meier survival curves.

#### Power calculation methods

Power calculations were carried out using the PS sample size program [21]. Conditional power at the interim analysis was computed using the method described in Jitlal et al. [20]. Estimates of loss of power due to the use of a non-binding conditional power futility boundary were computed via a simulation of 10,000 replications of a clinical trial with the null and alternative hypotheses as specified in the above power tables. For the simulated power calculations we assume an interim analysis at the 50% accrual time, and stopping if the probability of a statistically significant result (two-sided p-value < 0.05) is below 15%, based on a conditional power calculation [20].

#### 6.2 Data Security

and e for Treatment of Data will be entered into electronic case report forms (eCRFs) through OnCore® which is the Cancer Institute's clinical trials management system. These eCRFs are used to record subject data generated by subject events: typically labs, study medication administration or procedures of the protocol. Each user accesses the software using his/her Rutgers Net ID and password. Users are given access or permission to various areas of OnCore® based on their role within the Cancer Institute (I.e., data entry, regulatory, study coordination). Audit trails are built into the software to track when data entry was started, when the form was declared complete, when the form was monitored/queried, amended, and then finalized. OnCore® also functions as an honest broker and has the capability to provide deidentified data reports to the principal investigator or designee for analysis.

# 6.3 Data and Safety Monitoring

# A. Data/Safety Monitoring Plan

The Principal Investigator will be responsible for monitoring the data, assuring protocol compliance, and conducting the safety reviews at the specified frequency, which must be conducted at a minimum of once a month (including when re-approval of the protocol is sought). The Rutgers Cancer Institute of New Jersey's Human Research Oversight Committee (HROC) will be the DSMB of record. During the review process, the principal investigators (serving as monitor) will evaluate whether the study should continue unchanged, require modification/amendment, or close to enrollment. Either principal investigator, IRB or either Data or Safety Monitoring Committee have the authority to stop or suspend the study or require modifications at each institution. The PIs will be responsible for sharing this information in a timely fashion and coordinating appropriate parallel actions at the other institution.

An audit will be conducted following enrollment of the first two (2) or three (3) patients. Subsequent audits will occur dependent on the rate of enrollment by each participating site. More frequent audits of patient data and study conduct will occur if necessary. Prior audit findings and/or situations that may arise during the study will determine the need for more frequent auditing. All audit findings will be discussed with the principal investigator and report the HROC and the Rutgers University IRB.

# B. Data/Safety Monitoring Board Details



#### 6.4 Reporting Results

#### A. Individual Subjects' Results

Results of individual patient assessments will be shared with the individual patient as these are part of the medical record and impact medical care. These results are part of routine care (safety labs, routine radiology procedures, and physical examinations).

B. Aggregate Results Aggregate research results will not be shared with the study participants.

C. Professional Reporting

I

H

S

J

a

D. Clinical Trials Registration, Results Reporting and Consent Posting
ClinicalTrials.Gov Registration and Data Reporting: Under the terms of the Food and Drug
Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments
Act (FDAA), the Sponsor of the trial is solely responsible for determining whether the trial and its
results are subject to the requirements for submission to the Clinical Trials Data Bank,
<a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>. Information posted will allow subjects to identify potentially
appropriate trials for their disease conditions and pursue participation by calling a central contact
number for further information on appropriate trial locations and trial site contact information.

This is a research study which prospectively assigns human participants to health related interventions. The study will be registered on clinicaltrials.gov per FDA Regulations within 21 days of enrollment of the first participant and updated at least every 6 month.

6.5 Secondary Use of the Data N/A

7.0 Research Repositories – Specimens and/or Data

8.0 Approvals/Authorizations

9.0 Bibliography

 Lai CC, Shih TP, Ko WC, Tang HJ, Hsueh PR. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges. Int J Antimicrob Agents. 2020 Feb 17:105924. doi: 10.1016/j.ijantimicag.2020.105924. [Epub ahead of print].

- 2. Wang LS, Wang YR, Ye DW, Liu QQ. A review of the 2019 Novel Coronavirus (COVID-19) based on current evidence. Int J Antimicrob Agents. 2020 [Epub ahead of print].
- WHO Director-General's opening remarks at media briefing on COVID-19 11 March 2020. [https://www.who.int/dg/speeches/detail/who-director-general-s-opening-remarks-at-the media-briefing-on-covid-19-11-march-2020]
- Wu Z, McGoogan JM. Characteristics of an important lesion from the coronavirus disease 2019 (COVID-19) outbreak in China: summary of a report of 72,314 cases from the Chinese Center for Disease Control and Prevention. JAMA. 2020 Feb 24. Doi: 10.1001/jama.2020.2648. [Epub ahead of print].
- 5. Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, et al. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res 2020; 10-0282.
- Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends 2020 Feb 19. Doi: 10.5582/bst.20202.0147. [Epub ahead of print].
- 7. Chinese Clinical Trial Registry. http://www.chictr.org.cn.
- Zhonghua Jie He Hu Xi Za Zhi. Multicenter collaboration group of Department of Science and Technology of Guangdong Province and Health Commission of Guangdong Province for chloroquine in the treatment of novel coronavirus pneumonia. Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia]. 2020 Mar 12; 43 (3):185-188. doi:10.3760/cma.j.issn.1001-0939.2020.03.009.
- Gautret P, Lagier J-C, Parola P, et al. Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. *Int. J. Antimicrob Agents* 105949 (2020) doi: 10.1016/j.ijantimicag.2020.105949.
- Biot C, Daher W, Chavain N, Fandeur T, Khalife J, Dive D, et al. Design and synthesis of hydroxyferroquinederivatives with antimalarial and antiviral activities. J Med Chem 2006; 49:2845-2849.
- Marmor MF, Kellner U, Lai TY, Melles RB, Mieler WF. American Academy of Ophthalmology. Recommendations on Screening for Chloroquine and Hydroxychloroquine Retinopathy (2016 Revision). Ophthalmology. 2016 Jun; 123(6):1386-94. doi: 10.1016/j.ophtha.2016.01.058. Epub 2016 Mar16.
- Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, et al. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Mar 9. pii: ciaa237. doi: 10.1093/cid/ciaa237. [Epub ahead of print].
- Raoult D, Houpikian P, Tissot Dupont H, Riss JM, Arditi-Djiane J, Brouqui P. Treatment of Q fever endocarditis: comparison of 2 regimens containing doxycycline and ofloxacin or hydroxychloroguine. Arch Intern Med. 1999 Jan25; 159 (2):167-73.





- 14. Lagier JC, Raoult D. Whipple's disease and Tropheryma whipplei infections: when to suspect them and how to diagnose and treat them. Curr Opin Infect Dis. 2018Dec; 31(6):463-470. doi: 10.1097/QCO.000000000000489. [x] Expert consensus on chloroquine phosphate for the treatment of novel coronavirus pneumonia.
- Armstrong N, Richez M, Raoult D, Chabriere E. Simultaneous UHPLC-UV analysis of hydroxychloroquine, minocycline and doxycycline from serum samples for the therapeutic drug monitoring of Q fever and Whipple's disease. J. Chromatogr. B Analyt. Technol. Biomed. Life Sci. 2017: 1060, 166-172.
- Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, et al. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 11. pii: S0140-6736(20)30566-3. doi: 10.1016/S0140-6736(20)30566-3. [Epub ahead of print].
- Retallack H, Di Lullo E, Arias C, Knopp KA, Laurie MT, Sandoval-Espinosa C, et al. Zika virus cell tropism in the developing human brain and inhibition by azithromycin. Proc Natl Acad Sci USA. 2016 Dec 13; 113 (50): 14408-14413. Epub 2016 Nov 29.
- Bosseboeuf E, Aubry M, Nhan T, de Pina, JJ, Rolain JM, Raoult D, et al. Azithromycin inhibits the replication of Zika virus. J Antivirals Antiretrovirals. 2018 10(1):6-11. doi: 10.4172/1948-5964.1000173.
- Bacharier LB, Guilbert TW, Mauger DT, Boehmer S, Beigelman A, Fitzpatrick AM, et al. Early administration of azithromycin and prevention of severe lower respiratory tract illnesses in preschool children with a history of such illnesses: A randomized clinical trial. JAMA. 2015 Nov 17; 314(19):2034-2044. doi:10.1001/jama.2015.13896.
- Jitlal M, Khan I, Lee SM, & Hackshaw, A. Stopping clinical trials early for futility: retrospective analysis of several randomized clinical studies. *Br. J. Cancer* 107, 910-917 (2012). http://dx.doi.org/10/1038%Fbjc.2012.344.
- 21. Dupont, WD & Plummer Jr., WD. Power and sample size calculations: A review and computer program. Control Clin Trials 11, 116-128 (1990). <a href="http://dx.doi.org/10.1016%2F0197-2456(90)90005-M">http://dx.doi.org/10.1016%2F0197-2456(90)90005-M</a>
- 23. Woosley, R. L., Heise, C. W., Gallo, T., Tate, J., Woosley, D., & Romero, K. A. (2013). QTdrugs List. Retrieved May 7, 2020, from www.CredibleMeds.org

| Appendix | A _ ( | Study | Flow | Table |
|-----------|-------|-------|------|-------|
| Appelluix | A 1 | Study | LINA | Iduic |

| Appendix A – Procedures | Screening<br>Day 0 <sup>4</sup> | D1 | D2 | D3 | D4 | D5 | D6 | D7 | D8 | D9 | D10 | D11-<br>D20 | Weekly<br>FUP x<br>4 <sup>2</sup> | Monthly<br>FUP x 6 <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed consent | X | | | | | | | | | | | | | |
| Baseline Medical<br>History | X | | | | | | | | | | | | | |
| Physical assessment | X | | | X | | | х | | | | Х | | | |
| Demographics | Х | | | | | | | | | | | | | |
| Electrocardiogram | Х | | | | | | | | | | | | | |
| CBCD, CRP, Ferritin,<br>D-Dimer, LDH and<br>Troponin | X | | | | | | x | | | | × | | | |
| Serum pregnancy (if applicable) | Х | | | | | | | | | | | | | |
| Eligibility Review | Х | | | | | | | | | | | | | |
| Randomization | Х | | | | | | | | | | | | | |
| Study Drug<br>Dispensing | Х | | | | | | X1 | | | | | | | |
| Azithromycin (Arm<br>1) | | Х | Х | X | X | X | | | | | | | | |
| Hydroxychloroquine sulfate (Arm 1 & 2) | | Х | Х | X | X | X | X | X | X | Х | X | | | |
| Placebo/<br>Hydroxychloroquine<br>sulfate (Arm 3) <sup>1</sup> | | Х | Х | Х | X | X | X | X | X | X | X | X | | |
| Research Blood<br>draw | х | | | X | | | Х | | | | | | | |
| Saliva, Oropharynx swabs | х | | | Х | | | Х | | | | | | | |
| Pill Diary Review | X | Х | Х | X | Х | X | X | X | X | X | X | Х | | |
| Daily Temperature<br>Review | X | X | Х | Х | Х | Х | X | X | X | X | X | X | X | X |
| Adverse Event<br>Review | | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | Х | X | X |
| Concomitant<br>Medication Review | Х | Х | Х | X | Х | X | Х | Х | X | Х | X | Х | | |
| COVID-19 Symptom<br>Questionnaire | X | X | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | X | X |
| Record other SOC<br>Procedures | X | Х | Х | Х | X | X | X | X | Х | Х | X | X | X | X |

- 1. Treatment will be administered Day 6 to D15 for Arm 3.
- 2. Phone assessments weekly x 4 weeks (+/- one day).
- 3. Phone assessments monthly x 6 months (+/- one week).
- 4. Screening and Day 1 visits may be combined. All procedures may be completed within 24 hours of screening visit.

Appendix B
Drugs associated with a known or possible risk of QT prolongation

| Drug class | Known risk | Possible risk |
|---|---|---|
| ADHD | | Atomoxetine |
| Alpha-blocker | | Alfuzosin |
| Analgesic | | Hydrocodone-ER<br>Tramadol |
| Anesthetic, general | Propofol<br>Sevoflurane | |
| Anti-androgen | | Degarelix<br>Leuprolide |
| Antianginal | Bepridil | |
| Antiarrhythmic | Amiodarone Disopyramide Dofetilide Dronedarone Flecainide Ibutilide Procainamide Quinidine Sotalol | |
| Antibiotic | Azithromycin Clarithromycin Erythromycin Ciprofloxacin Levofloxacin Moxifloxacin | Bedaquiline Gemifloxacin Norfloxacin Ofloxacin Telavancin Telithromycin Lefamulin |
| Anticancer | Arsenic trioxide<br>Vandetanib<br>Cesium Chloride | Encorafenib Toremifene Dpirubicin Fluorouracil (5-FU) Oxaliplatin Inotuzumab ozogamicin Glasdegib Midostaurin Ribociclib Tamoxifen Eribulin mesylate Lapatinib Osimertinib Capecitabine Sunitinib Bosutinib Dasatinib Nilotinib Bendamustine |

| Drug class | Known risk | Possible risk |
|---|---|---|
| | | Sorafenib Ceritinib Entrectinib Necitumumab Cobimetinib Dabrafenib Vemurafenib Tipiracil/Trifluridine Crizotinib Cabozantinib Pazopanib Lenvatinib Vorinostat Tazemetostat Romidepsin Vorinostat Panobinostat Ivosidenib Apalutamide Bortezomib |
| Anticoagulant | | Betrixaban |
| Anticonvulsant | | Ezogabine<br>Felbamate |
| Antidepressant, SNRI | | Venlafaxine |
| Antidepressant, SSRI | Citalopram<br>Escitalopram | Clomipramine<br>Lithium |
| Antidepressant, Tetracyclic | | Meprotiline Mirtazapine Desipramine Imipramine Nortriptyline Trimipramine |
| Antiemetic | Ondansetron<br>Droperidol<br>Chlorpromazine | Dolasetron<br>Granisteron<br>Palonosetron<br>Promethazine |
| Antifungal | Fluconazole<br>Pentamidine | |
| Antihypertensive | | Isradipine<br>Moexipril/hydrochlorothiazide<br>Nicardipine |
| Antimalarial | Chloroquine<br>Hydroxycholorquine | Artenimol/piperaquine<br>Artemether/Lumefantrine |
| Antimanic | | Lithium |

| Drug class | Known risk | Possible risk |
|---|---|---|
| Antineoplastic | | Giltertinib |
| Antipsychotics | Droperidol<br>Chlorpromazine<br>Haloperidol<br>Pimozide<br>Thioridazine | Perphenazine Promethazine Pimavanserin Asenapine Clozapine Iloperidone Lumateperone Paliperidone Lurasidone Aripiprazole |
| Antisense oligonucleotide | | Nusinersen |
| Antitubercular | | Pretomanid |
| Antiviral | | Efavirenz<br>Lopinavir/Ritonavir<br>Rilpivirine<br>Saquinavir |
| Antispasmodic | | Mirabegron |
| Cholinesterase inhibitor | Donepezil | |
| Dopamine agonist | | Apomorphine |
| Estrogen agonist/antagonist | | Toremifene |
| Glucosylceramide synthase inhibitor | | Eliglustat |
| Gonadotropin receptor agonist/antagonist | | Leuprolide |
| Gonadotropin-releasing hormone agonist/antagonist | | Degarelix |
| Histamine H <sub>2</sub> receptor antagonist | | Famotidine |
| Histamine 3 antagonist/inverse | | Pitolisant (Tiprolisant) |
| mmunosuppressant | | Tacrolimus |
| maging contrast agent | | Perflutren lipid microspheres |
| llicit drugs | Cocaine | |
| Muscle relaxants | | Tizanidine<br>Tolterodine |
| NMDA receptor antagonist | | Memantine |
| CNS Stimulant | | Atomoxetine |
| Dxytocic | | Oxytocin |
| Opiates | Methadone | Buprenorphine |
| Phosphodiesterase 3 inhibitors | Anagrelide<br>Cilostazol | |

| Drug class | Known risk | Possible risk |
|---|---|---|
| Phosphodiesterase 5 inhibitors | | Vardenafil |
| Progesterone antagonist | | Mifepristone |
| Sedative | | Dexmedetomidine |
| Somatostatin analog | | Pasireotide |
| Sphingosine phosphate receptor modulator | | Fingolimod |
| Unknown | | Dextromethorphan/Quinidine |
| Vasodilator, Coronary | Papaverine HCL (Intracoronary) | |
| Vesicular monamine transporter 2 inhibitor | | Deutetrabenazine |
| Vesicular monamine transporter 2 inhibitor | | Valbenazine |
| Vesicular monamine transporter 2 inhibitor | | Tetrabenazine |



Appendix C

# CINJ 002011 COVID-19 Baseline Questionnaire

| Are you complet | ting this Baseline Questionnaire online or in person at Online |
|---|---|
| a study site? | and a second describing of in personal E |
| a staay site: | In person at study site |
| Please indicate i | if you have been diagnosed with or treated for one or more of the following conditions: |
| | Diabetes mellitus |
| | High blood pressure or hypertension |
| | Asthma |
| | Chronic bronchitis, emphysema, or chronic obstructive pulmonary disease (COPD) |
| | Another chronic lung disease (specify ): |
| | Coronary artery disease, peripheral artery disease, angina, or heart attack (myocardial infarction) |
| | Congestive heart failure |
| | Stroke or transient ischemic attack (TIA) |
| | Atrial fibrillation |
| | Cancer other than non-melanoma skin cancer |
| | Chronic kidney disease (CKD) |
| | Crohn's disease, ulcerative colitis, or inflammatory bowel disease (IBD) |
| | Rheumatoid arthritis (RA), psoriasis, systemic lupus, multiple sclerosis, or another disorder |
| | for which you take medicine to lower your immune system (immunosuppressant) |
| Please write the | names of all the medicines you have taken in the last week, including over-the-counter medicine |
| supplements, pro | |
| Medicine 1 | Medicine 8 |
| Medicine 2 | Medicine 9 |
| Medicine 3 | Medicine 10 |
| Medicine 4 | Medicine 11 |
| Medicine 5 | Medicine 12 |
| Medicine 6 | Medicine 13 |
| | Medicine 14 |

List any other medicines you take here, separated by commas.



| 是是大型技术,所是这些企业的技术是自然 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Do you ever take a probiotic? 0, 1 | Never | | | | | | | | |
| 1,0 | Occasionally | , such | n as wh | nen I tak | e anti | biotic | s or h | nave dia | rrhea |
| | es, regularly | | | | | | | | |
| Have you ever received pneumococcal vaccines | 20052 | | neumo | ovax-23 | )? | | | 0, No | |
| | | | | | | | H | 1.0000000000000000000000000000000000000 | |
| | | | | | | | H | 1, Yes | |
| Did you receive the influenza vaccine this past s | 2 | | | | | | Ц | 2, I do | n't know |
| bid you receive the initidenza vaccine this past's | easonr | | | 0, No | | | | | |
| | | | | 1, Yes | | | | | |
| S DE N SET SER N D SE | | | Ш | 2, I do | n't kn | ow | | | |
| In the last week, have you had a new fever > 10 | 0° F? | | | 0, No | | | | | |
| | | | | 1, Yes | | | | | |
| | | | П | | | | ut die | d not ta | ke my |
| In the last week, have you had a new cough? | | | _ | tempe | erature | ∍. | | | |
| in the last week, have you had a new cough? | L | | ), No | | | | | | |
| Table Table of Land Co. | | mmd . | ., Yes | | | _ | | 7038 | |
| In the last week, have you felt new shortness of | breath or h | ad ne | ew diffi | iculty bi | reathir | ng? | | | 0, No |
| | | | | | | | | | 1, Yes |
| In the last week, have you had new vomiting? | | ] 0 | , No | | | | | | |
| | | | , Yes | | | | | | |
| In the last week, have you had new diarrhea (m | ultiple wate | ry sto | ools)? | | | 0, No | ) | | |
| | | | | | | 1, Ye | S | | |
| In the last week, have you had a new loss of sme | ell or taste? | | | | | 0, No | ) | | |
| | | | | | | 1, Ye | S | | |
| Indicate when you have lost your sense of smell | , taste, or be | oth. | | | | 0, Sm | nell | | |
| | | | | | П | 1, Ta | ste | | |
| | | | | | | 2, Bo | th sn | nell and | taste |
| In the last week, have you received care or beer for coronavirus in an office or clinic? | tested [ | ] 0 | , No | | _ | | | | |
| and the state of t | | ] 1 | , Yes, f | or one | or mor | e of t | he al | oove syr | mptoms |
| | г | 7 2 | . Yes, f | or anot | her re | ason | | | |
| What diagnosis (or diagnoses) were you given? | | | | | | | | | |
| PARTIES THE STATE OF THE STATE | ¥ | | | | | | | | |

| Name of emergency contact: | |
|---|---|
| Relationship of emergency contact: | <ul> <li>O, Spouse/Partner</li> <li>1, Child</li> <li>2, Parent</li> <li>3, Sibling</li> <li>4, Grandparent</li> <li>5, Aunt</li> <li>6, Uncle</li> <li>7, Cousin</li> <li>8, Unrelated Adult/Roommate</li> <li>9, Friend</li> <li>10, Neighbor</li> <li>11, Other (specify below)</li> </ul> |
| Mobile phone number of emergency contact: | |
| Relationship of second emergency contact: | 0, Spouse/Partner 1, Child |

ycin and quine for Treatment of

| Mobile phone number of second emergency contact: | | |
|---|---|---|
| How would you describe your ethnicity? | | 1, Hispanic, Latino, Latina, or Latinx |
| 200 | | 2, Middle Eastern or North African descent |
| | | 0, None of the above |
| | | 3, Prefer not to report |
| How would you describe your race? | | 1, American Indian or Alaskan Native |
| | | 2, Asian |
| | | 3, Black or African American |
| | | 4, First Nations, Inuit, or Métis |
| | | 5, Native Hawaiian or other Pacific Islander |
| | | 0, White |
| | | 6, Other |
| | П | 7, Prefer not to report |



# Appendix D

# CINJ 002011 COVID-19 Follow-up Questionnaire

| Day: | Patient: | | | | 11.2 | | 11 |
|---|---|---|---|---|---|---|---|
| Update on how you are feeling | | | | | | | |
| In the last day, have you had a new feve | .00° F? | | | 0, No | | | |
| | | | | 1, Yes | | | |
| | | | | 1, I felt feverish but did not take my temperature. | | | |
| In the last day, have you had a new cough? | | | 0, No | | | | |
| | | | 1, Yes | | | | |
| In the last day, have you felt new shortness | of breath or ha | ad no | ew diffic | ulty breathing | 15 | | 0, No |
| | | | | | | | 1, Yes |
| In the last day, have you had new vomiting? | | | 0, No | | | | |
| | | | 1, Yes | | | | |
| In the last day, have you had new diarrhea (I | multiple water | y sto | ools)? | | 0, No | | |
| | | | | | 1, Yes | | |
| In the last day, have you had a new loss of sr | nell or taste? | | | | 0, No | | |
| | | | | | 1, Yes | | |
| Indicate when you have lost your sense of smell, taste, or both. | | | • | | 0, Smell | | |
| | | | | | 1, Taste | | |
| | | | | | 2, Both sı | mell and | taste |
| In the last day, have you had any additional symptoms? | | | | | 0, No | | |
| | | | | | 1, Yes | | |
| In the last day, have you taken any new med | | 0, No | | | | | |
| If so please list below | | | | | 1, Yes | | |

| In the last day, have you receive office or clinic? | are or had tests in ar | | 0, No | | |
|---|---|---|---|---|---|
| | | | 1, Yes | | |
| Document test or procedures | | | | | |
| | | | | *************************************** | *************************************** |
| Please provide all temperatures | AM: | | | | |
| recorded on your log in the last 24 hours. | Mid day. | | | | |
| 24 110015. | Mid-day: | | | | |
| | Afternoon: | | | | |
| | Night: | | | | |
| | Might. | | | | *************************************** |
| In the last day, have you taken you as prescribed? | ır study medication | | 0, No | | |
| | | | 1, Yes | | |
| | | Ш | | | |